CLINICAL TRIAL: NCT00399230
Title: A Comparison of Optive in Patients Previously Using Systane for the Treatment of Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 5279
Record Dates: First submitted 2006-11-09; First posted 2006-11-14 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

INTERVENTIONS:
Drug: Optive

SUMMARY:
To evaluate the effectiveness of NGT (Optive) vs. Systane Tears for patients with moderate to severe dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* · Dry eye disease diagnosis

  * Patients must currently be using Systane tears at least once a day and for at least 1 month.
  * Normal lid position and closure
  * Male or female of legal age of consent
  * Informed consent has been obtained
  * Likely to complete all required follow-up visits

Exclusion Criteria:

* · Concurrent enrollment in an investigational drug or device study, or participation in such a study within 30 days of entry into this study.

  * Subject has a condition, or is in a situation which, in the investigator's opinion, may put the subject at a significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Rajpal, MD, Principal Investigator — See Clearly Vision Group
Locations (1):
- Dr. Rajpal, McLean, Virginia, United States